CLINICAL TRIAL: NCT01786694
Title: Feasibility of Microdialysis by Laparoscopy
Acronym: MTM-COLON-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI2012_843_0022; 2012-A01218-35 (Other: ID-RCB)
Record Dates: First submitted 2013-02-01; First posted 2013-02-08 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Rectal Cancer
Keywords: rectum; microdialysis; quality of life
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cma microdialysis catheter placement (Experimental): At the end of the surgery the cma microdialysis catheter is placed near the anastomosis
  Interventions: Device: cma microdialysis catheter placement

INTERVENTIONS:
Device: cma microdialysis catheter placement — the microdialysis catheters are sold by CMA

SUMMARY:
The aim of this pilot study is to evaluate the feasibility of microdialysis by laparoscopy in order to identify anastomotic leaks after rectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* rectal disease requiring proctectomy with anastomosis and stomy
* proctectomy by laparoscopy
* written consent

Exclusion Criteria:

* history of colorectal surgery
* rectal surgery without anastomosis
* breastfeeding or pregnancy
* ASA score IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
functional success of microdialysis | postoperative day 5
  the functional success of microdialysis is defined as abnormal values localised at the microdialysis catheter

SECONDARY OUTCOMES:
anastomotic leaks rate | postoperative day 30
  the anastomotic leaks rate is defined as the number of anastomotic leaks validated by a CT scan
superficial surgical site infection rate | postoperative day 30
  the surgical site infection rate is defined as the number of infection near the incision
the mortality rate | postoperative day 30
  the mortality rate is defined as the number of death after the surgery
the quality of life after the surgery | postoperative day 30
  the quality of life will be evaluated with the QLQ C30 CR 29 prior to the surgery, at the hospital discharge and on postoperative day 30

CONTACTS AND LOCATIONS:
Overall Officials: jean marc regimbeau, MD, PhD, Principal Investigator — CHU amiens
Locations (1):
- Amiens University Hospital, Amiens, France

REFERENCES:
- [Background] Hogberg N, Carlsson PO, Hillered L, Meurling S, Stenback A. Intestinal ischemia measured by intraluminal microdialysis. Scand J Clin Lab Invest. 2012 Feb;72(1):59-66. doi: 10.3109/00365513.2011.629307. Epub 2011 Nov 21. PMID 22103734
- [Background] Deeba S, Corcoles EP, Hanna GB, Pareskevas P, Aziz O, Boutelle MG, Darzi A. Use of rapid sampling microdialysis for intraoperative monitoring of bowel ischemia. Dis Colon Rectum. 2008 Sep;51(9):1408-13. doi: 10.1007/s10350-008-9375-4. Epub 2008 May 24. PMID 18500500
- [Background] Verdant CL, Chierego M, De Moor V, Chamlou R, Creteur J, de Dieu Mutijima J, Loi P, Gelin M, Gullo A, Vincent JL, De Backer D. Prediction of postoperative complications after urgent laparotomy by intraperitoneal microdialysis: A pilot study. Ann Surg. 2006 Dec;244(6):994-1002. doi: 10.1097/01.sla.0000225092.45734.e6. PMID 17122625